CLINICAL TRIAL: NCT01786421
Title: Observational Study of Diurnal Triglyceridemia in Relation to Alcohol Intake
Brief Title: Diurnal Triglyceridemia in Relation to Alcohol Intake
Status: Completed | Type: Observational
Sponsor: Sint Franciscus Gasthuis (Other)
Responsible Party: Principal Investigator, Ana Torres do Rego, Medical Doctor, Sint Franciscus Gasthuis
Other Study IDs: AlcoholTG_SFG_2013
Record Dates: First submitted 2013-01-29; First posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Healthy Subjects; Hyperlipidemias; Type 2 Diabetes Mellitus; Cardiovascular Diseases
Keywords: Ethanol; Lipemia; Postprandial; Triglyceride
MeSH Terms: conditions — Hyperlipidemias; Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- General population: Healthy volunteers,patients with hyperlipidemia,a known medical history of cardiovascular diseases or type 2 diabetes mellitus.

SUMMARY:
The purpose of this study is to determine the impact of alcohol consumption in diurnal triglyceridemia in a free living situation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Patients with:

* Hyperlipidemia
* Type 2 Diabetes Mellitus
* Cardiovascular diseases

Exclusion Criteria:

* Renal disease
* Liver disease
* Thyroid disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were healthy volunteers or patients with hyperlipidemia or a known medical history of cardiovascular diseases, type 2 diabetes mellitus participating in several clinical studies with the same protocol, aimed to investigate factors influencing postprandial lipemia
Sampling Method: Probability Sample
Enrollment: 273 (Actual)
Dates: Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Determination of diurnal triglyceridemia depend on alcohol intake | For 3 days.
  Capillary triglyceridemia was measured by a triglyceride testing device on six fixed time-points.

SECONDARY OUTCOMES:
Gender differences in diurnal triglyceridemia by alcohol consumption | For 3 days

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Sint Franciscus Gasthuis, Rotterdam, Rotterdam
  - Utrecht University Medical Center, Utrecht, Utrecht